CLINICAL TRIAL: NCT02539303
Title: In-vivo Demineralization of Calcific Peripheral Arterial Disease (PAD) Using Local Delivery of Yamani-15/5 Chemical Solution
Brief Title: Delivery of Yamani-15/5 Chemical Solution for PAD
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to enroll subjects
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Houssam Farres, M.D., Dr. Houssam Farres, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-001279
Record Dates: First submitted 2015-08-27; First posted 2015-09-03 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Infusion of Yamani-15/5 chemical solution.
  Interventions: Drug: Yamani-15/5 chemical solution

INTERVENTIONS:
Drug: Yamani-15/5 chemical solution — A 20 ml of Yamani-15/5 will be directly infused into the diseased (calcific) arterial distribution.

SUMMARY:
This is a feasibility pilot study to evaluate the impact of local delivery of Yamani-15/5 (combination of L-Lactic acid 15% and D-Gluconic acid 5%) on vascular calcification of lower extremities in patients with severe peripheral arterial disease (PAD) who were deemed to have unreconstructable arterial disease and who have already been scheduled to undergo limb amputation (below knee or above knee amputation).

ELIGIBILITY:
Subject has severe calcific PAD who have been deemed to have unreconstructable arterial disease and who have already been scheduled to undergo limb amputation (below knee or above knee amputation).

Exclusion:

* Patients who will be undergoing amputation of the limb because of infection, osteomyelitis or cancer.
* Patients with chronic kidney disease stage V (unless on dialysis).
* Patients with liver cirrhosis.
* Patients with history of deep vein thrombosis or pulmonary embolization in the last 3 months.
* Patients with history of stroke in the last 3 months.
* Patients with unstable angina or history of myocardial infarction in the last 3 months.
* Patients with sepsis, respiratory failure, hypovolemic shock or cardiogenic shock.
* Women who are pregnant or nursing.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2022-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Feasibility | Change from baseline
  Percent of arterial lumen patency measured by angiography and compared to baseline.

SECONDARY OUTCOMES:
Safety as measured by the number of participants with treatment-related adverse events as assessed by Common Toxicity Criteria for Adverse Effects v4.0. | Compared to baseline
  Number of participants with treatment-related adverse events as assessed by Common Toxicity Criteria for Adverse Effects v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Houssam Farres, MD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials